CLINICAL TRIAL: NCT00231751
Title: The Malmö International Brother Study (MIBS)
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Other Study IDs: MIBS
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2005-10-04 (Estimated); Status verified 2005-09

CONDITIONS: Hemophilia A With Inhibitors
Keywords: Hemophilia A; Inhibitors
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Existing data support the concept that a genetic predisposition for inhibitor development exists. The aim of the Malmö International Brother Study (MIBS) is to evaluate genetic factors associated with the development of inhibitory antibodies in patients with hemophilia.

DETAILED DESCRIPTION:
Inhibitory antibodies to factor VIII develop in 10-15% of all patients with hemophilia A and in 25-30% of patients with the severe form of the disease after exposure to factor VIII concentrates. Both genetic and environmental risk factors for inhibitor development have been evaluated, but in most cases without consistent results. Among the genetic factors, an association between large rearrangements of the factor VIII and IX genes and a higher risk for inhibitors has been described. However, a majority of patients with null mutations, including the intron 22 inversion, do not develop inhibitory antibodies. It is obvious that other genetic markers influencing the immune response to replacement therapy in patients with hemophilia remain to be identified and the aim of Malmö International Brother Study (MIBS) is to characterize these factors.

ELIGIBILITY:
Inclusion Criteria:

-Mild, moderate or severe hemophilia A or B and one or more brothers with mild, moderate or severe hemophilia A or B

Exclusion Criteria:

-Absence of sufficient information to classify inhibitor status

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-11; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Jan Astermark, M.D., Ph.D., Principal Investigator — Skane University Hospital
Locations (1):
- Malmö University Hospital, Malmo, Sweden

REFERENCES:
- [Background] Astermark J, Oldenburg J, Escobar M, White GC 2nd, Berntorp E; Malmo International Brother Study study group. The Malmo International Brother Study (MIBS). Genetic defects and inhibitor development in siblings with severe hemophilia A. Haematologica. 2005 Jul;90(7):924-31. PMID 15996930
- [Background] Astermark J, Berntorp E, White GC, Kroner BL; MIBS Study Group. The Malmo International Brother Study (MIBS): further support for genetic predisposition to inhibitor development in hemophilia patients. Haemophilia. 2001 May;7(3):267-72. doi: 10.1046/j.1365-2516.2001.00510.x. PMID 11380630
- [Background] Astermark J, Berntorp E. Malmo International Brother Study (MIBS): an international survey of brother pairs with haemophilia. Vox Sang. 1999;77 Suppl 1:80-2. doi: 10.1159/000056723. PMID 10529695
- [Derived] Astermark J, Donfield SM, Gomperts ED, Schwarz J, Menius ED, Pavlova A, Oldenburg J, Kessing B, DiMichele DM, Shapiro AD, Winkler CA, Berntorp E; Hemophilia Inhibitor Genetics Study (HIGS) Combined Cohort. The polygenic nature of inhibitors in hemophilia A: results from the Hemophilia Inhibitor Genetics Study (HIGS) Combined Cohort. Blood. 2013 Feb 21;121(8):1446-54. doi: 10.1182/blood-2012-06-434803. Epub 2012 Dec 6. PMID 23223434